CLINICAL TRIAL: NCT06178302
Title: DEscripitive Patient Analysis to Enable Risk-based Quality Improvement Measures in a lArge iNternal mediCIne grouP Practice - The EMANCIPATE Study
Brief Title: DEscripitive Patient Analysis to Enable Risk-based Quality Improvement Measures in a lArge iNternal mediCIne grouP Practice
Acronym: EMANCIPATE
Status: Not yet recruiting | Type: Observational
Sponsor: Imed19 (Other)
Responsible Party: Sponsor
Other Study IDs: Imed19 EMANCIPATE2023
Record Dates: First submitted 2023-12-03; First posted 2023-12-20 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Liver Dysfunction; Thyroid; Atherosclerosis; Heart Failure; Intestinal Disease; Heart Diseases
MeSH Terms: conditions — Liver Diseases; Thyroid Diseases; Atherosclerosis; Heart Failure; Intestinal Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Clinical trials often include patients from large hospitals or university clinics. Information on patients cared for at offices from statutory health insurance-accredited physicians represent evidence gaps.

Aims/Objectives:

The present study has three aims: First, to systematically describe the patient population of a large group practice for internal medicine. Second, to identify high-risk patients using established risk scores. And third, to include routine imaging data to optimize patient management.

Methods/Facility Enrolling Participants: This is a prospective, observational study assessing patients' baseline characteristics, risk evaluation and integrating data from imaging test. The setting of the present study is a large group practice for internal medicine which consists of statutory health insurance-accredited physicians. Study participants will be included during daily routine, real-world clinical care and therefore represent all-comers fulfilling the inclusion criteria:

1. Female or male patients aged above 18 years diagnosed with chronic liver disease, undergo on-site endoscopy, suffer from atherosclerosis, heart failure, are diagnosed with abnormal serum thyroid-stimulating hormone (TSH) levels, either overt or latent hypo- or hyperthyroidism, or are diagnosed with solitary or multiple thyroid nodules.
2. Routine laboratory results available within the last 3 months.
3. Available imaging data within the last 3 months performed on site. Perspective: The study is designed to evaluate the current situation and quality of health care in defined patient populations in the routine clinical setting of a large-scale public office. These data will provide a profound rationale to identify quality issues and limitations in our performance of guideline-conform treatment in routine patient care.

ELIGIBILITY:
1. Female or male patients aged above 18 years diagnosed with chronic liver disease, undergo on-site endoscopy, suffer from atherosclerosis, heart failure, are diagnosed with abnormal serum thyroid-stimulating hormone (TSH) levels, either overt or latent hypo- or hyperthyroidism, or are diagnosed with solitary or multiple thyroid nodules.
2. Routine laboratory results available within the last 3 months.
3. Available imaging data within the last 3 months performed on site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population of a large group practice for internal medicine
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristics | Baseline/time of study inclusion
  To describe the baseline characteristics (age, weight, height, routinely assesses laboratory parameters such as creatinin, thyroid hormones, liver enzymes, lipids) of patients with heart failure in a community based internal medicine practice.
Risk evaluation | At baseline and as available during routine clinical follow-up, up to 10 years (no formal follow-up visits/time frames))
  Describe risk according to risk scores (the CHADS-VASC Score, the EU- TIRADS score, the ASCVD risk score, FIB-4 Score )
Quality of care evaluation | At baseline and as available during routine clinical follow-up, up to 10 years (no formal follow-up visits/time frames)
  Describe achievement of individual treatment targets according to current guidelines (Lipid targets, bloodpressure targets)

IPD SHARING:
Plan to Share IPD: Undecided